CLINICAL TRIAL: NCT01196949
Title: The Effectiveness of Combined Manipulation and Rehabilitation Versus Rehabilitation Only, in the Management of Chronic Ankle Instability
Brief Title: Comparing Manipulation and Rehabilitation to Rehabilitation Only, in the Management of Chronic Ankle Instability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cleveland Chiropractic College (Other)
Collaborators: Durban University of Technology (Other)
Responsible Party: James W. Brantingham, Cleveland Chiropractic College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCC08132010A
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2010-09-27 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Ankle Instability
Keywords: Ankle; Chronic; Instability; Manipulative; Rehabilitative; Manipulation; Rehabilitation
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manipulative and Rehabilitative Therapy (Active Comparator)
  Interventions: Other: Manipulative and Rehabilitative Therapy
- Rehabilitative Therapy (Active Comparator)
  Interventions: Other: Rehabilitative Therapy

INTERVENTIONS:
Other: Manipulative and Rehabilitative Therapy — Participants will receive 6 treatments over a 3 to 5 week time frame. A minimum of one day and maximum of 3 days between treatments. This group will receive high velocity low amplitude thrust to a minimum of 1 and maximum of 3 restricted segments within the mortise joint, subtalar joint and tarsal along with the same rehabilitation protocol as the other group.
  Arms: Manipulative and Rehabilitative Therapy
Other: Rehabilitative Therapy — Participants will receive education and training in the home exercises. This group is only required to attend the treatment facility for outcome measure readings and if they have any questions about the research protocol or check if they are performing their exercises correctly. A Theraband will be utilized for the peroneal muscle strengthening; 3 sets of 12 repetitions. Proprioception will be conducted on a Bosu Ball; 10 minutes per period. This protocol will be conducted everyday at home for the 5 week study. A diary will be required to record compliance and indicate how exercises should be performed.
  Arms: Rehabilitative Therapy

SUMMARY:
It is hypothesized that a combination approach would produce increased clinically and statistically significant outcomes as opposed to standard single intervention, inclusive of comparatively greater reduction in pain, improvement in range of motion, proprioception and function with an associated quicker recovery time.

Chronic ankle instability (CAI) is a frequently encountered condition of the musculoskeletal system. Various individual treatment options have previously been compared to one another in clinical trials, however there is paucity of literature with regards to combined treatment choices versus individual therapy. The purpose of this study is to investigate the relative effectiveness of combined manipulation and rehabilitation versus rehabilitation only, in the management of CAI.

The study will be conducted as a single blinded randomised and comparative clinical trial at Cleveland Chiropractic College and Durban University of Technology.

DETAILED DESCRIPTION:
Rationale

1. Inversion ankle sprains are the most frequently encountered injury to the ankle (Ferran and Maffulli, 2006) especially in the realm of the sporting arena (Balint et al, 2003; Delahunt, 2007; Bozzelle and Kishner, 2008). Up to 40 % of these acutely injured participants will progress to a state of chronic ankle instability (CAI) (Verhagen et al, 1995; Balint et al, 2003; Ajis and Maffulli, 2006; Ajis et al, 2006). Therefore the lateral ankle as well as the management of CAI requires further investigation with regard to treatment options.
2. Peroneal muscle weaknesses as well as proprioceptive deficits have been universally encountered in cases of CAI (Reid, 1992; Delahunt, 2007). Studies have indicated that coupled peroneal muscle strengthening and proprioception training of the ankle are seen as the most efficient means of rehabilitation for CAI (Reid, 1992; Ajis et al, 2006; Ajis and Maffulli, 2006; McBride and Ramamurthy, 2006; Caulfield, 2007; Lee and Lin, 2008). Pellow and Brantingham, (2001) and Gillman, (2004) have reported that manipulation is also a successful intervention tool for the treatment of CAI, documenting a statistically significant reduction in pain (p=0.007), improved range of motion (p=0.199) in the ankle joint as well as improved general functioning of the ankle (p=0.004). It has been identified that there are three components (Richie, 2001; Sefton et al, 2008) that contribute to the persistence of CAI namely joint fixations (in the mortise and subtalar joint) as well as muscular (Richie, 2001) and proprioceptive alterations (Richie, 2001; Delahunt, 2007).
3. It is hypothesised that a combination approach would produce increased clinically and statistically significant outcomes as opposed to standard single intervention, inclusive of comparatively greater reduction in pain, improvement in range of motion, proprioception and function with an associated quicker recovery time (Green et al, 2001; Eisenhart et al, 2003; Collins,2004; Vicenzino et al, 2006). There are insufficient studies, particularly high quality studies, with the required methodology, to make a definitive decision regarding whether this is supported (Van der Wees et al, 2006; Whitman et al, 2009). Additionally chiropractors will typically manage a participant with CAI with a combination of manipulation and rehabilitation, at present no research using such combined therapy by chiropractors has yet been published (Brantingham et al, 2009).

3. Research Problem and Aims The aim of the study is to investigate the relative effectiveness of a combination of manipulation and rehabilitation as compared to rehabilitation only in the treatment for CAI, in terms of participantive and objective clinical assessments.

The specific objectives of the study are:

1. To determine the relative effectiveness of manipulation and rehabilitation versus rehabilitation only, to the ankle joint in terms of objective assessments (algometer, berg balance scale, weight bearing ankle dorsiflexion test and foot and ankle disability index in participants experiencing CAI syndrome).
2. To determine the relative effectiveness of manipulation and rehabilitation versus rehabilitation only, to the ankle joint in terms of participantive assessments (visual analogue scale and motion palpation) in participants experiencing CAI syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with grade one (Grade I: evidence of minimal swelling with minimal dysfunction, point tenderness over joint, absence of positive anterior drawers sign) or grade two (Grade II: moderate amount of swelling and haemorrhage over the ankle with pain more do on weight bearing). Potentially positive anterior drawers sign but with no varus laxity CLAI (Reid, 1992; Pellow and Brantingham, 2001; Rimando, 2008).
2. Participants between the ages of 18 - 45 years (Pellow and Brantingham, 2001; Chowdry et al, 2003; Parker, 2005).
3. Participants that are clinically diagnosed as having CLAI: the presence of 4 or more of a combination of symptoms including lateral ankle pain, joint weakness, oedema (Tatro-Adams et al, 1995), joint crepitus, adhesions resulting in the formation of fixations in the joint and ligamentous laxity (Reid, 1992; Pellow and Brantingham, 2001; Ajis and Maffulli, 2006; McBride and Ramamurthy, 2006; Caulfield, 2007).
4. Participants with a visual analogue scale (vas) (Liggins, 1982; Salaffi et al, 2003) score of between 20 and 70 millimetres to maintain homogeneity within the sample (Mouton, 1996).
5. Participants with a foot/ankle disability Index (FADI) (Hale and Hertel, 2005) of between 50 and 90 to maintain homogeneity within the sample (Mouton, 1996).
6. Participants with a berg balance scale (Kornetti et al, 2004) of less than 45/56 to maintain homogeneity within the sample (Mouton, 1996).
7. Participants must have the presence of fixations in either the mortise joint, the subtalar joint or the tarsals (Brantingham et al, 2007).
8. Participants that give informed consent to participate in the research.
9. Participants on muscle relaxants or any anti inflammatory medication will be required to have a wash out period of three days before participating in the study (Poul et al, 1993; Seth, 1999).

Exclusion Criteria:

1. Participants who have experienced an acute injury or acute re-injury (prior to or during the study) will be excluded from the study because it does not comply with the six-week interval (i.e. chronic injuries) (Pellow and Brantingham, 2001).
2. Participants with balance disorders of a neurological and/or otological and/or vascular cause of dizziness that may mimic instability and defective proprioception at the ankle level (Clark and Burden, 2005; Kynsberg et al, 2006).
3. Participants with connective tissue disorders that create excessive generalised ligamentous laxity, participants with these conditions will not benefit from the treatment with generalised hyper laxity of ligaments.
4. Participants with grade three CAI/ gross mechanical instability of the lateral ankle complex as the severity of this grade of injury usually requires surgical intervention and is unresponsive to conservative therapy (Reid, 1992; Pellow and Brantingham, 2001; Rimando, 2008).Grade III: severe swelling and haemorrhage with positive anterior drawers sign and rupture of ligamentous structures.
5. Participants that are contraindicated to adjustments, which include but may not be limited to (Kirkaldy - Willis and Burton, 1992).

Absolute contraindications, Destructive injury of the skeletal structures of the body; fractures and dislocations of all varieties; neurological damage as in Cauda equina syndrome, abdominal aortic aneurysm, referred pain of a visceral nature.

Relative Contraindications, bone demineralization, psychosomatic conditions, anticoagulant therapy and/or conditions where hemorrhaging may be present and Spondyloarthropathies.

Participants with secondary manifestations of any of the following conditions, which may compromise balance/ proprioception, which are contraindicated to rehabilitation, which include and may not be limited to (Frontera, 1999).

Dizziness that is present during the treatment Peripheral vascular disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-10 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 3months
  Gold standard subjective pain scale

SECONDARY OUTCOMES:
Foot Ankle Disability Index | 3 months
  General Ankle Function Assessment Tool

CONTACTS AND LOCATIONS:
Overall Officials: James W Brantingham, Dc, PhD, Principal Investigator — Cleveland Chiropractic College; Danella Lubbe, Principal Investigator — Durban University of Technology
Locations (1):
- Durban University of Technology, Durban, South Africa

REFERENCES:
- [Background] Ferran NA, Maffulli N. Epidemiology of sprains of the lateral ankle ligament complex. Foot Ankle Clin. 2006 Sep;11(3):659-62. doi: 10.1016/j.fcl.2006.07.002. PMID 16971255
- [Background] Balint GP, Korda J, Hangody L, Balint PV. Regional musculoskeletal conditions: foot and ankle disorders. Best Pract Res Clin Rheumatol. 2003 Feb;17(1):87-111. doi: 10.1016/s1521-6942(02)00103-1. PMID 12659823
- [Background] Delahunt, E. 2007. Neuromuscular contributions to functional instability of the ankle joint. Journal of Bodywork and Movement Therapies, 11:203-213.
- [Background] Bozzelle, J.R. and Kishner, S. Recurrent Ankle Sprains. [Online] Available: http://emedicine.com, [Accessed August 2009].
- [Background] Ajis A, Maffulli N. Conservative management of chronic ankle instability. Foot Ankle Clin. 2006 Sep;11(3):531-7. doi: 10.1016/j.fcl.2006.07.004. PMID 16971246
- [Background] Reid, C.D. 1992. Sports Injury Assessment and Rehabilitation. United States of America: Churchill Livingston Inc
- [Background] McBride DJ, Ramamurthy C. Chronic ankle instability: management of chronic lateral ligamentous dysfunction and the varus tibiotalar joint. Foot Ankle Clin. 2006 Sep;11(3):607-23. doi: 10.1016/j.fcl.2006.07.009. PMID 16971252
- [Background] Caulfield, B. 2000. Functional Instability of the Ankle Joint, features and underlying causes. Physiotherapy, 86:8
- [Background] Lee AJ, Lin WH. Twelve-week biomechanical ankle platform system training on postural stability and ankle proprioception in subjects with unilateral functional ankle instability. Clin Biomech (Bristol). 2008 Oct;23(8):1065-72. doi: 10.1016/j.clinbiomech.2008.04.013. Epub 2008 Jul 14. PMID 18621453
- [Background] Pellow JE, Brantingham JW. The efficacy of adjusting the ankle in the treatment of subacute and chronic grade I and grade II ankle inversion sprains. J Manipulative Physiol Ther. 2001 Jan;24(1):17-24. doi: 10.1067/mmt.2001.112015. PMID 11174691
- [Background] Green T, Refshauge K, Crosbie J, Adams R. A randomized controlled trial of a passive accessory joint mobilization on acute ankle inversion sprains. Phys Ther. 2001 Apr;81(4):984-94. PMID 11276181
- [Background] van der Wees PJ, Lenssen AF, Hendriks EJ, Stomp DJ, Dekker J, de Bie RA. Effectiveness of exercise therapy and manual mobilisation in ankle sprain and functional instability: a systematic review. Aust J Physiother. 2006;52(1):27-37. doi: 10.1016/s0004-9514(06)70059-9. PMID 16515420
- [Background] Brantingham JW, Globe G, Pollard H, Hicks M, Korporaal C, Hoskins W. Manipulative therapy for lower extremity conditions: expansion of literature review. J Manipulative Physiol Ther. 2009 Jan;32(1):53-71. doi: 10.1016/j.jmpt.2008.09.013. PMID 19121464